CLINICAL TRIAL: NCT02654366
Title: Social Network Intervention for Syringe Exchange Registrants
Brief Title: Community Supported Risk Reduction for Syringe Exchange Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00080615; 1R34DA040507-01 (NIH)
Record Dates: First submitted 2015-09-25; First posted 2016-01-13 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Substance Use Disorders; Risk Reduction
Keywords: Syringe exchange; HIV risk reduction; Drug-free community support
MeSH Terms: conditions — Substance-Related Disorders; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Supported Risk Reduction Group (Experimental): Six weekly sessions will be scheduled during daytime and evening hours to accommodate the daily schedules of BNEP registrants and their CSPs. Each session meets for 60 minutes. Groups will consist of 5-6 BNEP registrant-CSP dyads (10-12 individuals). While BNEP registrants and CSPs attending the group together will receive an attendance incentive, BNEP registrants attending without a CSP will not earn one. The group leader will follow a manual that includes a structured outline. The group manual content combines risk reduction / treatment readiness and community outreach approaches. Following the introduction, each group session is divided into two components: 1) Risk Reduction and Treatment Readiness (30 min) and 2) Community Outreach skills (20 min).
  Interventions: Behavioral: Risk Reduction Group

INTERVENTIONS:
Behavioral: Risk Reduction Group — The Risk Reduction and Treatment Readiness skills component includes six modules: 1) BNEP services and substance abuse treatment; 2) nature of chemical dependence (severity/chronicity and medical aspects); 3) infectious diseases (HIV and Hepatitis C virus (HCV) information); 4) injection drug use risk reduction (effective equipment cleaning and drug-splitting techniques); 5) sex risk reduction (reducing high-risk behaviors and effective condom use); and 6) overdose prevention.
  The Community Outreach skills component is devoted to discussing the benefits of recovery-focused social support, and directing BNEP registrants and their CSPs to participate in activities together (as determined in the group session) at least 1 time per week to work toward expanding the scope of drug-free social support.

SUMMARY:
Efforts to help syringe exchange registrants employ additional HIV risk reduction strategies are often thwarted by strong social networks that reinforce substance use and other risky injection use and sexual behaviors. The proposed study addresses this important problem by evaluating the feasibility and efficacy of a novel Community Supported Risk Reduction group. This structured intervention works with injection drug users and at least one drug-free family or friend to mobilize social support, teach HIV risk reduction skills, develop treatment readiness, and support participation in community activities designed to expand drug-free social networks.

DETAILED DESCRIPTION:
Participants of syringe exchange programs routinely suffer from untreated or under-treated substance use disorder, a situation that is associated with significant individual and public health costs. These individuals are also routinely embedded within social networks that reinforce continued drug use and related HIV-risk behaviors. The welfare of these individuals and the public's health can be improved by interventions directed toward reducing drug use risks and expanding drug-free support . Previous work by the investigators has demonstrated that an intervention combining an HIV risk reduction/treatment readiness group with behavioral contingencies is highly associated with increased rates of treatment enrollment and re-engagement, and reduced rates of drug use and HIV-injection risks, for up to one year. This protocol extends this work by adding a new component to the HIV risk reduction/treatment readiness group designed to expand social support and facilitate social network change. This intervention requires syringe exchange registrants to attend the group with a drug-free family or friend from their personal network that can provide stable support and encourage harm reduction and treatment seeking. This intervention uses an alteration network change model and posits that repeated exposure to drug-free community support collaterally reduces exposure to network members that support risk behaviors. This model also provides a pathway to modifying existing social networks by facilitating interaction with the personal social networks of drug-free family and friends. The intervention is supported by research showing that substance users report substantial pockets of drug-free family or friends in their social networks. It is also supported by community reinforcement principles that have shown efficacy in treatment samples, but have not been applied to out-of-treatment drug users. The present study has four primary aims. The first is to characterize natural drug-free support in the social networks of syringe exchangers. The second is to develop a Community Supported Risk Reduction group for syringe exchange participants and their community support. This group teaches skills for HIV risk reduction, treatment seeking, and healthy network expansion. The third and fourth aims are to obtain new data on the feasibility and efficacy of this intervention. Primary outcomes include changes in: 1) perceived social support, and 2) HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria (for Baltimore Needle Exchange Program registrants):

* Baltimore Needle Exchange Program (BNEP) registration
* Injection heroin use
* Identifies a drug-free community support person (CSP)
* Not currently receiving substance abuse treatment

Exclusion Criteria (for BNEP registrants):

* Pregnancy
* Acute medical problem that requires urgent medical management
* Presence of a thought disorder, delusions, hallucinations, or imminent risk of harm to self or others
* Unable to read

Exclusion Criteria (for CSPs):

* Submission of a drug-positive urine sample
* Pregnancy
* Acute medical problem that requires urgent medical management
* Presence of a thought disorder, delusions, hallucinations, or imminent risk of harm to self or others
* Unable to read

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Perceived social support as assessed by the QRI "support" scale | Monthly for 3 months
  The investigators anticipate that Baltimore Needle Exchange Program (BNEP) registrants will demonstrate greater levels of perceived social support (QRI "support" scale, a continuous measure) across follow-ups (compared to baseline). Mixed model analyses will be used to evaluate change from baseline to follow-up measures (Months 1, 2, 3). The two remaining QRI subscales ("conflict"; "depth") will also be examined using a similar analytic approach.
HIV drug risk behaviors as assessed by the Risk Behavior Survey | Monthly for 3 months
  The investigators anticipate that BNEP registrants will have lower rates of any drug use risk behaviors (Risk Behavior Survey) across the 3-month evaluation compared to baseline. Drug use risks include any use of a used needle, cooker and cotton for injection or splitting drugs. Generalized Estimating Equations (GEE) will be used to assess change from baseline to follow-up measures (Months 1, 2, 3).
HIV sex risk behaviors as assessed by the Risk Behavior Survey | Monthly for 3 months
  Changes in any sex risk behaviors (Risk Behavior Survey) will be examined using Generalized Estimating Equations (GEE) to assess change from baseline to follow-up measures (Months 1, 2, 3). The investigators expect significant reductions only for the subset of individuals including a romantic partner as a Community Support Person (CSP).

SECONDARY OUTCOMES:
Number of participants enrolled in substance abuse treatment | Monthly for 3 months
  Following each group session, BNEP registrants interested in enrolling in substance abuse treatment will have an opportunity to schedule a referral to a treatment program. Substance abuse treatment enrollment (including treatment name, modality, start date, stop date, days in treatment) will be assessed at months 1, 2, 3 using a series of questions in the Risk Behaviors Survey.
Rates of injection drug use | Monthly for 3 months
  The Drug Use, Injection, and Sexual Risk Behaviors Survey will be administered at months 1, 2, and 3 to assess rates of injection drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kidorf, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No